CLINICAL TRIAL: NCT06920953
Title: A Prospective Observational Study to Evaluate Participant Satisfaction and Quality of Life With Catheter Washouts in Adults Living With Long-Term Catheters and Currently Using Uro-Tainer® Polihexanide 0.02%
Brief Title: Participant Satisfaction and Quality of Life With Catheter Washouts in Adults Living With Long-Term Catheters and Currently Using Uro-Tainer® Polihexanide 0.02%
Acronym: UTP Washout
Status: Not yet recruiting | Type: Observational
Sponsor: B. Braun Ltd. Centre of Excellence Infection Control (Industry)
Responsible Party: Sponsor
Other Study IDs: BA-O-H-24092
Record Dates: First submitted 2025-03-25; First posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Catheter Associated Urinary Tract Infection
Keywords: Catheter Washouts; Suprapubic long-term catheter

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Uro-Tainer® Polihexanide 0.02% (acronym: UTP washout) is a sterile, single-use, water-based solution (100 ml) currently used in clinical practice in the UK (and Europe) for the irrigation of Long-Term-Catheter. This medical device is intended for the maintenance of indwelling urethral and suprapubic Long-Term-Catheter to aid removal of deposits, tissue waste, clots, and mucus.

In this study of people living with Long-Term-Catheter and currently using UTP washouts as part of their standard clinical care, the following will be investigated :

* Participant satisfaction with their UTP washout
* Impact of UTP washout plan on their QoL
* Adverse events (blockage, SCAUTI, others)
* Participant adherence to their current washout frequency plan. This is an observational study. The participants are those currently using UTP washouts as prescribed by their clinical care team. There will be no change in treatment for study purposes.

DETAILED DESCRIPTION:
Several Long-Term-Catheter (LTC) washouts policies and maintenance solutions are used in clinical practice for prevention and/or management of LTC adverse events. Washouts used are of different types (normal saline, acidic, antimicrobial); volumes (50 ml, 2 x 30 ml, and 100 ml) and frequency of administration. The recent Cochrane review assessed the best available evidence and found insufficient evidence to determine whether prophylactic LTC washout policies had a beneficial or harmful effect on any of the outcomes in participants with LTC.

Most recently the CATHETER II RCT in the UK faced difficulties in recruitment and was terminated with 80 participants (target was 600). The RCT compared a policy of weekly prophylactic washout using either saline or acidic washouts to no washout policy. Despite the small sample size, there were trends towards lower rates of blockage and S-CAUTI in the groups using prophylactic washouts. The results did not reach statistical significance possibly due to the small sample size.

In-addition to the mechanical benefit of washouts such as the saline, antimicrobial washout solutions aim to reduce or prevent bacterial growth and reduce LTC blockages.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 years
* Participant is having a urethral or suprapubic long-term catheter (LTC) in situ for more than 28 days and no plan for discontinuation of LTC at the time of recruitment
* Currently using the LTC washout maintenance solution Uro-Tainer® Polihexanide 0.02%
* Able to undertake LTC washouts or has a designated person (relative, friend, other informal carer, or paid/NHS healthcare worker) able to perform washouts
* Able to complete the study documentation or has a designated person able to assist with study documentation
* Informed consent obtained

Exclusion Criteria:

* Age younger than 18 years
* Intermittent self catheterisation
* Pregnant or contemplating pregnancy or breastfeeding
* Ongoing S-CAUTI (until treatment is complete)
* Visible haematuria (unless investigated/treated)
* Known allergies to the LTC washout solution
* Current bladder cancer (until treatment is complete and participant discharged from cancer surveillance program)
* Known bladder stones (until treatment is complete)
* Not able to communicate or to give consent including participants with incapacity to consent
* Any other clinical and social reasons that would be deemed by the recruitment team to be unsuitable for the study
* Simultaneous participation in another clinical trial
* in case of hypersensitivity (allergy) to PHMB, chlorhexidine, or excipient of the solution.
* several days after surgery on the bladder or the urinary tract
* for open wounds, the inner and middle ear, the central nervous systems, eyes, hyaline cartilage, and meninges

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults (≥ 18 years) living in the community with urethral or suprapubic long-term (> 28 days) catheter (LTC) and currently undertaking Uro-Tainer® Polihexanide 0.02 % washouts
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Long-Term-Catheter participant satisfaction with their washout policy | At the end of the study (day 84)
  The participants' satisfaction with their washout is rated on the visual analogue scale "Participants" satisfaction with their washout solution - Uro-Tainer® Polihexanide 0.02%', with a minimum value of '0' and a maximum value of '10'. The minimum value means 'Not satisfied', the maximum value means 'Very satisfied'.

SECONDARY OUTCOMES:
Impact of washouts on participants QoL | At two visits (day 1 and day 84)
  Quality of Life assessed on ICIQ-LTCqol 12/12 (disease specific questionnaire), including
  * eight questions to the topic "Catheter function and concern", and to each question a VAS "How much does this bother you", with a value from 0 (= overall good) to 10 (= overall bad),
  * three questions to the topic "Lifestyle impact", and
  * four unscored questions, and to each question a VAS "How much does this bother you", with a value from 0 (= overall good) to 10 (= overall bad).
Impact of washouts on state of health | At two visits (day 1 and day 84)
  Quality of Life assessed with the questionnaire EQ-5D-5L, including fife questions, and EQ-5D-VAS "How good or bad your health is TODAY?", with a value from 0 (= The worst health you can imagine) to 100 (= The best health you can imagine.)
Adverse events: Long-Term-Catheter (LTC) blockage requiring an intervention; symptomatic LTC-related urinary tract infections (S-CAUTI) | At each visit (1-5), day 1 (baseline), day 21, day 42, day 63 and day 84 (close-out visit), and continuously between the visits, if an adverse event is reported by the participant.
  Lont-Term-Catheter washouts diary

IPD SHARING:
Plan to Share IPD: No